CLINICAL TRIAL: NCT03421873
Title: Effectiveness and Safety of a Clinical Assessment and 0h/1h Troponin Rule-Out Protocol
Acronym: ESC-TROP
Status: Completed | Type: Observational
Sponsor: Ulf Ekelund (Other)
Collaborators: Region Skane (Other); Lund University (Other)
Responsible Party: Sponsor-Investigator, Ulf Ekelund, Principal Investigator, Professor of Emergency Medicine, Region Skane
Organization: Region Skane (Other)
Other Study IDs: ESC-TROP20172018
Record Dates: First submitted 2018-01-21; First posted 2018-02-05 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Chest Pain; Acute Coronary Syndrome; Myocardial Infarction; Unstable Angina
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention (Implementation) group: Chest pain patients enrolled during a 10 month period after a change in routine care, i.e. the implementation of a 0h/1h hs-cTnT protocol
  Interventions: Other: 0h/1h hs-cTnT protocol
- Control group: Chest pain patients managed at the 3 intervention EDs during the corresponding 10 months of the previous year (intervention hospitals acting as their own controls) as well as chest pain patients managed during the corresponding before-and-after period at EDs not implementing the protocol (concurrent controls).

INTERVENTIONS:
Other: 0h/1h hs-cTnT protocol — Implementation of a 0h/1h hs-cTnT protocol in routine care
  Groups: Intervention (Implementation) group

SUMMARY:
Chest pain is a common presenting complaint at the Emergency Department (ED). Many of these patients undergo lengthy assessments in the ED or are admitted which contributes to ED and hospital crowding as well as a substantial health care burden. The now commonly used high-sensitivity cardiac troponin assays enable faster rule-out of acute myocardial infarction (AMI). The European Society of Cardiology (ESC) recommend the use of a 0h/1h high-sensitivity cardiac troponin T (hs-cTnT) protocol, but all studies so far have been observational. The safety and effectiveness of the protocol when implemented in routine care is thus unknown.

The aim of this study is to determine the safety and effectiveness of the ESC 0h/1h hs-cTnT protocol, supplemented with clinical assessment and ECG, when implemented in routine care.

DETAILED DESCRIPTION:
STUDY DESIGN:

ESC-TROP is a before-and-after implementation study with concurrent controls that will evaluate the safety and effectiveness of a 0h/1h hs-cTnT protocol. The intervention group will consist of ED chest pain patients enrolled during 10 months after implementation of this protocol in routine care at the three intervention sites, and the control groups will be chest pain patients managed at the same EDs during the corresponding 10 months of the previous year, as well as chest pain patients managed during the same before-and-after period at two EDs not implementing the protocol (concurrent controls).

OBJECTIVES:

To determine the safety and effectiveness of the ESC 0h/1h hs-cTnT protocol, supplemented with clinical assessment and ECG, when implemented in routine care.

ELIGIBILITY CRITERIA:

All patients with an ED visit with a primary complaint of non-traumatic chest pain will be identified through the electronic ED patient log and screened for eligibility.

IMPLEMENTED PROTOCOL:

ESC guidelines state that the 0h/1h hs-cTnT protocol should be used in conjunction with clinical assessment and the ECG, and these items are therefore incorporated in the protocol, which also reflects real-life practice. A 1h hs-cTnT is defined as a second hs-cTnT sample drawn 45 - 90 minutes from the sample at presentation (0h).

OUTCOMES:

Se outcomes section. Outcomes will be compared in the 10-month periods before and after the implementation at all five hospitals, and the differences in change will be compared between intervention and control hospitals.

FOLLOW-UP:

Follow-up will be performed using data from a comprehensive regional electronic patient record system as well as Swedish national registries.

DATA MANAGEMENT AND STATISTICAL ANALYSES:

Data management and statistical analyses will be performed by Clinical Studies Sweden, Forum South. For the primary safety outcome, event rate after implementation (intervention group) will be compared to event rate in the control period using a non-inferiority approach

SAMPLE SIZE:

If it is assumed that the event rate is 0.4% among discharged patients in the control period and 0.5% after implementation, 4396 discharged patients would be needed both before and after the implementation (i.e. a total of 8792) to statistically determine that the event rate after implementation is non-inferior to that in the control period, with a two-sided alpha risk of 0.05 and a power of 0.80. The non-inferiority margin has been set to 0.5 percentage units as there is consensus that a <1% incidence of AMI/death within 30 days represents good safety for a diagnostic strategy in chest pain patients.

Based on a total of 13100 annual chest pain patients at the three EDs and a 25% exclusion rate, a study period of 10 months will give enrollment of about 8200 patients. If 55% are discharged from the ED, about 4500 patients will be discharged both before and after implementation (i.e. a total of about 9000).

With this sample size, and an estimated median ED length of stay (LOS) in discharged patients in the control group of 240 minutes, it will be possible to detect a difference in ED LOS of about 14 minutes with a power of 0.80 and alpha of 0.05. This sample size will thereby provide adequate power to detect a clinically significant difference in ED LOS for the co-primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* ED presentation with a primary complaint of non-traumatic chest pain
* Age ≥18 years

Exclusion Criteria:

* A final diagnosis of STEMI during the index visit
* No hs-cTnT ordered
* Patient leaving against medical advice
* No Swedish personal identification number
* Previous enrollment
* Unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All ED patients with a primary complaint of chest pain will be screened for eligibility
Sampling Method: Probability Sample
Enrollment: 16000 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
AMI and all-cause death | 30 days from ED presentation
  Comparison of the rate of AMI and all-cause death within 30 days from ED presentation in patients discharged from the ED during the intervention period versus the control period (safety)
ED length of stay | Through discharge from the ED, on average 5 hours after ED presentation
  Comparison of ED length of stay in patients discharged from the ED during the intervention period versus the control period (effectiveness)

SECONDARY OUTCOMES:
Proportion of ED patients discharged | Through discharge from the ED, on average 5 hours after ED presentation
  Comparison of the proportion of patients discharged from the ED during the intervention period versus the control period
Proportion of patients fulfilling 0h/1h hs-cTnT criteria who have undergone objective testing | 30 days from ED presentation
  Proportion of patients fulfilling 0h/1h hs-cTnT criteria (0h hs-cTnT <5 ng/L or a 0h hs-cTnT <12 ng/L with a 1h increase <3 ng/L) who have undergone objective testing (exercise stress test, myocardial perfusion imaging, CT coronary angiography, coronary angiography) within 30 days during the intervention period.
Non-ACS coronary care unit admissions | Throughout index hospital visit, on average 2 days after ED presentation
  Comparison of the proportion of patients without acute coronary syndrome (ACS) admitted to the coronary care unit during the intervention period versus the control period.
Inappropriate coronary angiographies | Throughout index hospital visit, on average 2 days after ED presentation
  Comparison of the proportion of patients who undergo inappropriate coronary angiographies during the intervention period versus the control period
Total hospital length of stay | Through discharge from the index hospital visit, on average 2 days after ED presentation
  Comparison of total hospital length of stay during the intervention period versus the control period.
ED revisits | 30 days from ED presentation
  Comparison of the proportion of patients with 30-day ED revisits during the intervention period versus the control period.
New admissions | 30 days from ED presentation
  Comparison of the proportion of discharged patients with admissions to inpatient care within 30 days during the intervention period versus the control period.
Health care costs | 30 days from ED presentation
  Comparison of health care costs within 30 days during the intervention period versus the control period. These data will be presented in a separate sub-study.

CONTACTS AND LOCATIONS:
Overall Officials: Arash Mokhtari, MD, PhD, Principal Investigator — Lund University, Skåne University Hospital, Department of Internal and Emergency Medicine, Department of Cardiology, Lund, Sweden; Ulf Ekelund, MD, PhD, Principal Investigator — Lund University, Skåne University Hospital, Department of Internal and Emergency Medicine, Lund, Sweden
Locations (5):
- Sweden (5):
  - Helsingborg General Hospital, Helsingborg
  - Kristanstad Central Hospital, Kristianstad
  - Skåne University Hospital, Lund
  - Skåne University Hospital, Malmo
  - Ystad Hospital, Ystad

REFERENCES:
- [Derived] Mokhtari A, Forberg JL, Sandgren J, Hard Af Segerstad C, Ellehuus C, Ekstrom U, Bjork J, Lindahl B, Khoshnood A, Ekelund U. Effectiveness and Safety of the ESC-TROP (European Society of Cardiology 0h/1h Troponin Rule-Out Protocol) Trial. J Am Heart Assoc. 2024 Nov 5;13(21):e036307. doi: 10.1161/JAHA.124.036307. Epub 2024 Oct 29. PMID 39470043
- [Derived] Gilje P, Mohammad MA, Roos A, Ekelund U, Bjork J, Lindahl B, Holzmann M, Mokhtari A. A Single High-Sensitivity Cardiac Troponin T Strategy for Ruling Out Myocardial Infarction. Emerg Med Int. 2024 Mar 25;2024:2241528. doi: 10.1155/2024/2241528. eCollection 2024. PMID 38567081